CLINICAL TRIAL: NCT06205524
Title: An Exploratory, Randomized, Double-Blind, Dose-Ranging Study to Evaluate the Safety and Immunogenicity of TI-0010 Vaccine to Prevent COVID-19 Caused by SARS-CoV-2 in Healthy Adults Aged 18-59 Years
Brief Title: A Study to Evealuate Safety and Immunogenicity of TI-0010 SARS-CoV-2 Vaccine in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Drug Clinical Trial Institute of the Second Affiliated Hospital of Bengbu Medical College (Other)
Collaborators: Therorna (Industry)
Responsible Party: Principal Investigator, Xiaoli Li, an associate chief physician, National Drug Clinical Trial Institute of the Second Affiliated Hospital of Bengbu Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TI-0010-10102
Record Dates: First submitted 2023-12-18; First posted 2024-01-16 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: COVID-19; COVID-19 Immunisation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- cohort 1 (Experimental): Participants will receive 2 intramuscular (IM) injections of either TI-0010 or Placebo at Dose Level 1 on Day 0 and Day 28
  Interventions: Biological: TI-0010; Biological: Placebo
- cohort 2 (Experimental): Participants will receive 1 intramuscular (IM) injection of either TI-0010 or Placebo at Dose Level 1 on Day 0
  Interventions: Biological: TI-0010; Biological: Placebo
- cohort 3 (Experimental): Participants will receive 2 intramuscular (IM) injections of either TI-0010 or Placebo at Dose Level 2 on Day 0 and Day 28
  Interventions: Biological: TI-0010; Biological: Placebo
- cohort 4 (Experimental): Participants will receive 1 intramuscular (IM) injection of either TI-0010 or Placebo at Dose Level 2 on Day 0
  Interventions: Biological: TI-0010; Biological: Placebo

INTERVENTIONS:
Biological: TI-0010 — Sterile liquid for injection
Biological: Placebo — 0.9% sodium chloride (normal saline) injection

SUMMARY:
This study is a randomized, double-blind, placebo controlled clinical exploratory study to evaluate the safety, tolerability and immunogenicity of TI-0010 vaccine in healthy adults aged 18-59. TI-0010 was manufactured by Therorna Inc. TI-0010 is a novel lipid nanoparticles (LNP) -encapsulated circRNA-based vaccine targeting RBD of SARS-CoV-2. Up to one hundred subjects will be enrolled into one of 4 cohorts. Low-dose(Dose Level 1) is for Cohort 1 and Cohort 2 , and the high dose (Dose Level 2) for Cohort 3 and Cohort 4. Cohort 1 and Cohort 3 receive 2 doses (with a 28 day interval) via intramuscular injection respectively, and Cohort 2 and Cohort 4 receive 1 dose via intramuscular injection respectively. Participants are randomized to receive TI-0010 or placebo in a 4:1 ratio.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo controlled clinical exploratory study to evaluate the safety, tolerability and immunogenicity of TI-0010 vaccine in healthy adults aged 18-59. TI-0010 was manufactured by Therorna Inc. TI-0010 is a novel lipid nanoparticles (LNP) -encapsulated circRNA-based vaccine targeting RBD of SARS-CoV-2. Up to one hundred subjects will be enrolled into one of 4 cohorts. Low-dose(Dose Level 1) is for Cohort 1 and Cohort 2 , and the high dose(Dose Level 2) for Cohort 3 and Cohort 4. Cohort 1 and Cohort 3 receive 2 doses (with a 28 day interval) via intramuscular injection respectively, and Cohort 2 and Cohort 4 receive 1 dose via intramuscular injection respectively. Participants are randomized to receive TI-0010 or placebo in a 4:1 ratio. Follow-up visits will occur Days 3,7,14 and 28 post each vaccination, as well as 3, 6, 9 and 12 months for the single dose recipients after vaccination and for those who receive two doses post the second vaccination. The primary objective is to evaluate the safety and tolerability of the TI-0010 vaccine in adults within 28 days post each vaccination. The secondary objective is to evaluate the humoral and cellular immune responses of the TI-0010 vaccine in adults after a single dose or two doses of vaccination, to evaluate the safety of the TI-0010 vaccine within 1 year after vaccination in the adult population and to evaluate the immune persistence of TI-0010 vaccine after a single dose and two doses of administration.

ELIGIBILITY:
Inclusion Criteria:

* Understands and agrees to comply with the study procedures and provides written informed consent.
* Participant shall be in good general health within the age range of 18 to 59 years old when signing ICF, and can comply with study procedures
* For participant of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy after signing ICF, agreement to continue adequate contraception through 3 months following vaccine administration, and not currently breastfeeding.
* Participants have not received any SARS-CoV-2 vaccine before screening; Or if participants have previously received SARS-CoV-2 vaccination, who vaccinated at least 6 months from the last vaccination date.
* Participant has tested positive or had COVID-infection related symptoms at least 4 months prior to screening.

Exclusion Criteria:

* Arm 2/4 only: Individuals haven't completed full vaccination schedule with any approved or investigational COVID-19 vaccines.
* Individuals with clinically significant laboratory or ECG abnormalities at Screening.
* BMI >30 kg/m2 or <18 kg/m2
* Positive RT-PCR test for SARS-CoV-2 at the screening site
* Known exposure to someone with SARS-CoV-2 infection or COVID-19 in the past 5 days
* Postive test for HBsAg or HCV
* Participant is acutely ill 4 weeks prior to Day1, or feberile (body temperature no less than 37.3 Celcius 72 hours prior to or at Day 1
* Has received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to Screenin or is anticipating the need for immunosuppressive treatment at any time during participation in the study
* Participation in a study of investigational drug/device 30 days prior to Screening
* Individuals with a history of autoimmune disease or an active autoimmune disease requiring therapeutic intervention
* History of sever adverse reaction associated with a vaccine and/or severe allergic reaction to any component of the study intervention(s)
* Previous vaccination with any vaccine 28 days prior Screening
* Receipt of blood/plasma products or immunoglobulin 3 months prior Screening
* Other medical or psychiatric condition that may increase the risk of study participation or, in the investigator's judgment, make the individual inappropriate for the study

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
solicited adverse events (AEs) | Up to 14 days following each injection among all participants.
  solicited adverse events (AEs)
The incidence of abnormal changes in laboratory indicators (including blood routine, blood biochemistry, thyroid function, coagulation function, and urine routine. ) | Up to 3 days following each injection among all participants.
  The incidence of abnormal changes in laboratory indicators (including blood routine, blood biochemistry, thyroid function, coagulation function, and urine routine. )

SECONDARY OUTCOMES:
Geometric mean titer(GMT) of SARS-CoV-2 neutralizing antibodies | Baseline, 7 days, 14 days, 28 days after Dose 1； 7 days, 14 days, 28 days after Dose 2（only for Cohort 1/3）； 3 months, 6 months, 9 months and 12 months
  Geometric mean titer(GMT) of SARS-CoV-2 neutralizing antibodies
Geometric mean titer fold increase(GMI) of SARS-CoV-2 neutralizing antibodies compared to baseline | Baseline, 7 days, 14 days, 28 days after Dose 1； 7 days, 14 days, 28 days after Dose 2（only for Cohort 1/3）； 3 months, 6 months, 9 months and 12 months
  Geometric mean titer fold increase(GMI) of SARS-CoV-2 neutralizing antibodies compared to baseline
Seroconversion rates(SCRs) of SARS-CoV-2 neutralizing antibodies | Baseline, 7 days, 14 days, 28 days after Dose 1； 7 days, 14 days, 28 days after Dose 2（only for Cohort 1/3）； 3 months, 6 months, 9 months and 12 months
  Seroconversion rates(SCRs) of SARS-CoV-2 neutralizing antibodies
Geometric mean titer(GMT) of SARS-CoV-2 RBD-binding IgG | Baseline, 7 days, 14 days, 28 days after Dose 1； 7 days, 14 days, 28 days after Dose 2（only for Cohort 1/3）； 3 months, 6 months, 9 months and 12 months
  Geometric mean titer(GMT) of SARS-CoV-2 RBD-binding IgG
Geometric mean titer fold increase(GMI) of SARS-CoV-2 RBD-binding IgG compared to baseline | Baseline, 7 days, 14 days, 28 days after Dose 1； 7 days, 14 days, 28 days after Dose 2（only for Cohort 1/3）； 3 months, 6 months, 9 months and 12 months
  Geometric mean titer fold increase(GMI) of SARS-CoV-2 RBD-binding IgG compared to baseline
Seroconversion rates(SCRs) of SARS-CoV-2 RBD-binding IgG | Baseline, 7 days, 14 days, 28 days after Dose 1； 7 days, 14 days, 28 days after Dose 2（only for Cohort 1/3）； 3 months, 6 months, 9 months and 12 months
  Seroconversion rates(SCRs) of SARS-CoV-2 RBD-binding IgG
The ratio of IL-2, IL-4, IFN- γ and TNF- α in T lymphocyte subsets (CD4+，CD8+) and memory T cell subsets (CD4+，CD8+). | Baseline, 7 days, 14 days, 28 days after Dose 1； 7 days, 14 days, 28 days after Dose 2（only for Cohort 1/3）； 3 months, 6 months, 9 months and 12 months
  The ratio of IL-2, IL-4, IFN- γ and TNF- α in T lymphocyte subsets (CD4+，CD8+) and
Incidence of unsolicited Adverse Events (AEs) | From the time of first dose vaccination to day 28 after Dose 2 for Cohort 1/3; Up to day 28 after vaccination for Cohort 2/4.
  Incidence of unsolicited Adverse Events (AEs)
Incidence of Serious Adverse Events (SAEs), AE of Special Interest (AESIs), and Medically-attended Aes (MAAEs) | Day 0 to 12 months after Dose 2 for Cohort 1/3； Up to 12 months after vaccination for Cohort 2/4.
  Incidence of Serious Adverse Events (SAEs), AE of Special Interest (AESIs), and Medically-attended Aes (MAAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Li, Master, Principal Investigator — The Second Affiliated Hospital of Bengbu Medical College
Locations (1):
- The Second Affiliated Hospital Of BengBu Medical College, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available to other researchers